CLINICAL TRIAL: NCT00133471
Title: Evaluation of the Reactogenicity and Immunogenicity of Four Dosage Levels of Intramuscular Monovalent Inactivated Influenza A/H9N2 Vaccine With and Without MF59 Adjuvant in Ambulatory Adults
Brief Title: Inactivated Influenza A/H9N2 Vaccine With and Without MF59 Adjuvant in Ambulatory Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-019
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2009-01

CONDITIONS: Influenza
Keywords: Influenza, vaccine, A/H9N2, MF59, adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Group 1A: 3.75 mcg A/H9N2 no adjuvant (Experimental): 12 subjects to receive 3.75 mcg A/H9N2 with no adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine
- Group 2B: 7.5 mcg A/H9N2 plus MF59 adjuvant (Experimental): 12 subjects to receive 7.5 mcg A/H9N2 plus MF59 adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine; Drug: MF59 adjuvant
- Group 3A: 15 mcg A/H9N2 no adjuvant (Experimental): 12 subjects to receive 15 mcg A/H9N2 with no adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine
- Group 3B: 15 mcg A/H9N2 plus MF59 adjuvant (Experimental): 12 subjects to receive 15 mcg A/H9N2 plus MF59 adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine; Drug: MF59 adjuvant
- Group 4B: 30 mcg A/H9N2 plus MF59 adjuvant (Experimental): 12 subjects to receive 30 mcg A/H9N2 plus MF59 adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine; Drug: MF59 adjuvant
- Group 4A: 30 mcg A/H9N2 no adjuvant (Experimental): 12 subjects to receive 30 mcg A/H9N2 with no adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine
- Group 2A: 7.5 mcg A/H9N2 no adjuvant (Experimental): 12 subjects to receive 7.5 mcg A/H9N2 with no adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine
- Group 1B: 3.75 mcg A/H9N2 plus MF59 adjuvant (Experimental): 12 subjects to receive 3.75 mcg A/H9N2 plus MF59 adjuvant.
  Interventions: Biological: Influenza A/H9N2 vaccine; Drug: MF59 adjuvant

INTERVENTIONS:
Biological: Influenza A/H9N2 vaccine — A single lot of monovalent inactivated SA influenza A/H9N2 vaccine. All injections will be administered in a 0.5-mL volume into the deltoid muscle. Dosage levels are: 3.75-, 7.5-, 15-, and 30-mcg of HA of the vaccine strain with and without MF59 adjuvant.
Drug: MF59 adjuvant — MF59 adjuvant is an oil-in-water emulsion.
  Arms: Group 1B: 3.75 mcg A/H9N2 plus MF59 adjuvant; Group 2B: 7.5 mcg A/H9N2 plus MF59 adjuvant; Group 3B: 15 mcg A/H9N2 plus MF59 adjuvant; Group 4B: 30 mcg A/H9N2 plus MF59 adjuvant

SUMMARY:
The purpose of this study is to compare the body's reactions and immune responses after receiving different strengths of a H9N2 influenza virus vaccine with and without an adjuvant given into the arm muscle. Study participants will include up to 96 healthy adults, ages 18-34. The 4 dosages of the experimental H9N2 vaccine to be tested in this study are the following: 3.75, 7.5, 15, and 30-mcg (with and without MF59 adjuvant). Participants will be vaccinated on Days 0 and 28. Participants will record any vaccine side effects in a diary for 7 days following each vaccination. Participants will return to the clinic on days 2 and 7 after vaccination. Blood samples will be collected 7 days following each vaccination. Serum and nasal wash specimens will be collected before each vaccination and 4 weeks after injections (0, 4, and 8 weeks). Participants will be involved in study related procedures for up to 8 months.

DETAILED DESCRIPTION:
The primary goal of this study is to assess the safety of 4 different dosages of purified monovalent surface antigen (SA) influenza A/H9N2 virus vaccine with or without MF59 adjuvant and administered intramuscularly to ambulatory adults. The hypothesis is that all dosage levels of adjuvanted and nonadjuvanted vaccine will be well tolerated. The primary objective of this project is to evaluate the safety of 4 dosage levels of monovalent surface antigen (SA) influenza A/H9N2 virus vaccine given with or without MF59 adjuvant. The primary endpoint is the frequency and severity of solicited local and systemic adverse events in each vaccine dosage level group. The secondary objective of this project is to determine the immunogenicity of 4 dosage levels of monovalent surface antigen (SA) influenza A/H9N2 virus vaccine given with or without MF59 adjuvant. The secondary endpoints include the following: the proportions of subjects in each vaccine dosage group that achieve a serum HAI titer of at least 1:32 one month after the second vaccination; the geometric mean titer (GMT) of serum HAI antibody against the influenza A/H9N2 virus one month after the second vaccination; the rates of significant increases in titer between pre- and post-immunization serum samples (defined as seroconversion-i.e., increase in titer from <1:4 pre-immunization to at least 1:8 after vaccination, or 4-fold or greater increase in titer between pre- and post-immunization samples) 28 days after each vaccination (days 28 and 56); and the proportion of subjects with a 4-fold or greater increase in percent HA-specific antibody in nasal wash specimens for each vaccine group. The study will be a double-blind evaluation of 4 dosage levels of study vaccine. The 4 dosage levels to be tested are 3.75-, 7.5-, 15-, and 30-mcg of HA of the vaccine strain with and without MF59 adjuvant. Because all dosage levels are lower than the total hemagglutinin content of the FLUAD® vaccine used in Europe, subjects will be enrolled into all dosage and adjuvant groups concurrently using a randomized, double-blind study design. Ninety-six persons 18-34 years of age will be enrolled. A single lot of monovalent inactivated SA influenza A/H9N2 vaccine will be used throughout the trial. All injections will be administered in a 0.5-mL volume into the deltoid muscle. Screening and safety laboratory examinations will be assessed before the first dose and 7 days after each vaccination. Assessments for reactogenicity will be done for at least 20 minutes after each vaccination, in the clinic 2 and 7 days after each inoculation, via diary card for seven days after each vaccination, and via phone or other contact at 7 months after the first vaccination for any serious adverse events during the entire study period. Serum and nasal wash samples collected on days 0, 28, and 56 will be used to measure immunogenicity of the vaccine preparation. Participants will be involved in study related procedures for up to 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, healthy males and non-pregnant female adults 18-34 years of age.
* Able to give informed consent and available for all study visits.
* Able to understand and comply with planned study procedures.
* Women capable of bearing children must utilize an acceptable means of birth control (abstinence, oral contraceptives ("the pill"), intrauterine devices (IUDs), contraceptive implants under the skin, or contraceptive injections, or condoms with foam).
* On no concomitant medications except contraceptive medications.
* Normal screening laboratory values.

Exclusion Criteria:

* Known allergy to eggs or other components of vaccine.
* Prior receipt of an influenza A/H9N2 vaccine.
* Abnormal screening laboratory values (laboratory values must be within normal limits).
* Pregnancy, desire to become pregnant in the next 3 months, or lactation.
* Immunosuppression as a result of underlying illness or treatment.
* Use of oral or parenteral steroids, high-dose inhaled steroids (>800 mcg per day of beclomethasone dipropionate or equivalent), other immunosuppressive or cytotoxic drugs.
* Active neoplastic disease or history of any hematologic malignancy.
* Acute or chronic condition that (in the opinion of the investigator) would render vaccination unsafe or would interfere with the evaluation of responses (including but not limited to the following: known chronic liver disease, significant renal disease, unstable or progressive neurologic disorder, diabetes mellitus, transplant recipient).
* Use of experimental vaccines or medications within the month prior to study entry, or expected use of experimental or licensed vaccines or blood/blood products during the 1 month period after each inoculation with study vaccine.
* Receipt of immunoglobulin or other blood product within 3 months prior to enrollment.
* Receipt of other licensed vaccines within the preceding 2 weeks (inactivated vaccines) or 4 weeks (live vaccines).
* History of a severe reaction following vaccination with a contemporary influenza vaccine.
* Subject is enrolled in another clinical trial.
* Study personnel (those persons identified on study personnel logs).
* Any condition that in the opinion of the investigator would interfere with the interpretation or evaluation of the vaccine.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of solicited local and systemic adverse events in each vaccine dosage level group. | Duration of study.

SECONDARY OUTCOMES:
The proportions of subjects in each vaccine dosage group that achieve a serum HAI titer of at least 1:32. | One month after the second vaccination.
Rates of significant increases in titer between pre- and post-immunization serum samples 28 days after each vaccination. | Days 28 and 56.
The geometric mean titer (GMT) of serum HAI antibody against the influenza A/H9N2 virus. | One month after the second vaccination.
The proportion of subjects with a 4-fold or greater increase in percent HA-specific antibody in nasal wash specimens for each vaccine group. | Nasal wash samples collected on Days 0, 28, and 56.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Atmar RL, Keitel WA, Patel SM, Katz JM, She D, El Sahly H, Pompey J, Cate TR, Couch RB. Safety and immunogenicity of nonadjuvanted and MF59-adjuvanted influenza A/H9N2 vaccine preparations. Clin Infect Dis. 2006 Nov 1;43(9):1135-42. doi: 10.1086/508174. Epub 2006 Sep 25. PMID 17029131